CLINICAL TRIAL: NCT01895413
Title: Autologous Bone Marrow-derived Mesenchymal Stem Cells Used in the Treatment of Articular Cartilage Injury
Brief Title: Autologous Bone Marrow Mesenchymal Stem Cells Transplantation for Articular Cartilage Defects Repair
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexandra Cristina Senegaglia (Other)
Collaborators: Pontifícia Universidade Católica do Paraná (Other); Consultório Médico Dr. Alcy Vilas Boas Jr., Paraná, Brasil (Unknown); Hospital Marcelino Champagnat, Paraná, Brasil (Unknown); Fundação Araucária (Other)
Responsible Party: Sponsor-Investigator, Alexandra Cristina Senegaglia, PhD, Pontifícia Universidade Católica do Paraná
Organization: Pontifícia Universidade Católica do Paraná (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTM_LESÃO ARTICULAR-461/2010; CTM_LESÃO ARTICULAR-461/2010 (Other Grant/Funding Number: Fundação Araucária)
Record Dates: First submitted 2013-07-01; First posted 2013-07-10 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2015-10

CONDITIONS: Osteoarthritis
Keywords: Cartilage injury; Osteoarthritis; Mesenchymal stem cells
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal stem cells (Experimental): Bone marrow aspiration, Autologous bone marrow-derived mesenchymal stem cells
  Interventions: Procedure: Bone marrow aspiration

INTERVENTIONS:
Procedure: Bone marrow aspiration — Single intra-articular injection of autologous bone marrow-derived mesenchymal stem cells by arthroscopy

SUMMARY:
This is a non-randomized study aimed to determine the safety and efficacy of intra-articular injection of autologous bone marrow-derived mesenchymal stem cells in patients with knee articular cartilage defects.

DETAILED DESCRIPTION:
Osteoarthritis is the most prevalent joint disease, create articular cartilage defects is a frequent cause of joint pain, functional loss, and disability. Osteoarthritis often becomes chronic, and conventional treatments seek to ameliorate pain or improve mobility. However, these treatments rarely modify the course of the disease.Recent studies cell-based have shown encouraging results in both animal studies and a few human case reports. We designed a study to assess the safety and efficacy of osteoarthritis treatment with intra-articular injection of autologous bone marrow-derived mesenchymal stem cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with mild to moderate osteoarthritis (visual analogue scale)
* History of joint swelling, pain, stiffness, altered gait and loss of motion due to degenerative cartilage

Exclusion Criteria:

* Any past history of neoplasia and primary hematological disease
* Autoimmune disease or the medical history
* Systemic bone or cartilage disorders
* Acute or chronic communicable diseases including Hepatitis B, Hepatitis C and HIV
* Co-morbidity which the physician deems as a contraindication to stem cell transplantation and bone marrow biopsy
* Evidence of infection or fractures in or around the joint
* Contraindication to bone marrow aspiration
* Deviation from the axial axis (varus or valgus) greater than 12 degrees.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in WOMAC (Western Ontario and McMaster Universities)score | 3 months, 6 months, 9 months, 12 months

SECONDARY OUTCOMES:
Change from baseline in cartilage thickness at 6 months by MRI | 6 months
Knee pain relief (WOMAC and Lequesne scores) | 3 months, 6 months, 12 months
Change from baseline in progression of osteoarthritis at 12 months by plain radiograph (X-ray) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Brofman, PhD, Principal Investigator — Pontifícia Universidade Católica do Paraná
Locations (1):
- Centro de Tecnologia Celular, Pontifícia Universidade Católica do Paraná, Curitiba, Paraná, Brazil